CLINICAL TRIAL: NCT04515875
Title: Promoting Reengagement in Daily Meaningful Activity (PRIMA) Intervention for Adults With Mild Cognitive Impairment and Their Caregivers
Brief Title: PRIMA Intervention for Adults With Mild Cognitive Impairment and Their Caregivers
Acronym: PRIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Yvonne Lu, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IUPREMA0822; 1R01NR018162-01A1 (NIH)
Record Dates: First submitted 2020-06-15; First posted 2020-08-17 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment; Quality of life; Family caregivers
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The study conceptual framework is based on: 1) pilot work, 2) the Canadian Model of Occupational Performance that describes how individuals are motivated, adjust to psychosocial context and cognitive decline, and choose to participate in essential and meaningful daily activities; 3) problem-solving therapy principles. These frameworks, commonly applied to health problems in older populations, provide a systematic structure to improve task initiation and completion in adults with depression or executive dysfunction.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Following consent, the project manager will arrange a time convenient for patient-caregiver dyads to separately complete the baseline (T1) measures by phone. A data collector, blinded to randomization status, will administer all measures at all time points via phone interviews in a quiet, private setting and be available for questions following data collection. Immediately following completion of the T1 measures; and enter patient scores on the PHQ-9 depression scale directly to the database. A web-based computer-generated stratified randomization scheme will be used to assign the patient-caregiver dyads to DEMA or the information support group in 1:1 ratio using a block-randomized approach stratified on a depression score PHQ-9 ≤ 4 vs. PHQ-9 ≥ 5 or higher will be used to determine the randomization scheme. The Project Manager will immediately schedule Session 1. Only the statistician, PI, project manager, and the intervener will know the patient-caregiver dyad's randomization status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Engagement Meaningful Activity (DEMA) (Experimental): This group will receive 7 individualized sessions, 1 face-to-face session at week 1 and via 6 bi weekly telephone sessions delivered by a trained intervener. DEMA will use the principles of problem-solving therapy and consistent with the overall goals of this intervention; and will provide autonomy support, classify needs and goals, generalize manageable solutions, engage in self-selected activities under family support, and self-evaluate failure and success or renew problem-solving as needed. Each session consists: 1) MCI dyads are guided to use the principles of problem-solving therapy to review their personalized, self-selected meaningful activities and plan next steps to continue the activity, identify and establish a plan for additional activities; and 2) the intervener and dyad discuss one of the 6 topics in the Toolkit such as introducing of the intervention and meaningful activity concepts, understanding MCI, its treatments, management, resources, and planning for the future.
  Interventions: Behavioral: Daily Engagement Meaningful Activity (DEMA)
- Information Support (IS) (Placebo Comparator): This group will attend 1 face-to-face meetings to receive an overview of what will happen in the study and an initial Alzheimer disease educational brochure from the Alzheimer's Association (AA). The face-to-face sessions will take place at the IADC Clinical Core clinic, Indiana University Center of Excellence of Women's Health clinic, or Indiana School of Nursing conference room that based on patient-caregiver dyad's preference. Then they will receive 6 bi weekly follow-up phone calls and have the opportunity to ask only questions related to the educational materials. After completing Time 4 data collection, the patient-caregiver dyads will receive DEMA Self-Management Tool kit package through mail.
  Interventions: Behavioral: Information Support (IS)

INTERVENTIONS:
Behavioral: Daily Engagement Meaningful Activity (DEMA) — This group will receive 7 individualized sessions, 1 face-to-face session at week 1 and via 6 bi weekly telephone sessions delivered by a trained intervener. DEMA will use the principles of problem-solving therapy and consistent with the overall goals of this intervention; and will provide autonomy support, classify needs and goals, generalize manageable solutions, engage in self-selected activities under family support, and self-evaluate failure and success or renew problem-solving as needed. Each session consists: 1) MCI dyads are guided to use the principles of problem-solving therapy to review their personalized, self-selected meaningful activities and plan next steps to continue the activity, identify and establish a plan for additional activities; and 2) the intervener and dyad discuss one of the 6 topics in the Toolkit such as introducing of the intervention and meaningful activity concepts, understanding MCI, its treatments, management, resources, and planning for the future.
  Arms: Daily Engagement Meaningful Activity (DEMA)
Behavioral: Information Support (IS) — This group will attend 1 face-to-face meetings to receive an overview of what will happen in the study and an initial Alzheimer disease educational brochure from the Alzheimer's Association (AA). The face-to-face sessions will take place at the IADC Clinical Core clinic, Indiana University Center of Excellence of Women's Health clinic, or Indiana School of Nursing conference room that based on patient-caregiver dyad's preference. Then they will receive 6 bi weekly follow-up phone calls and have the opportunity to ask only questions related to the educational materials. After completing Time 4 data collection, the patient-caregiver dyads will receive DEMA Self-Management Tool kit package through mail.
  Arms: Information Support (IS)

SUMMARY:
The investigators developed and tested the Daily Engagement in Meaningful Activities (DEMA) intervention to improve life satisfaction and health outcomes for patients and caregivers. DEMA is a positive health focused, theoretically grounded, tailored, family-centered, multi-faceted intervention. Over 7 session, dyads work with a nurse to 1) identify meaningful activities, assess capacity, problem-solve barriers, and establish routines for engagement and 2) learn more about MCI by working through six Self-Management Toolkit topics (e.g., benefits of meaningful activity; planning the future). The investigators' purpose is to evaluate the efficacy of DEMA in a two-group randomized controlled trial with 200 patient/caregiver dyads (DEMA intervention vs. the information support (IS) attention control group).

DETAILED DESCRIPTION:
Approximately 20% of Americans over 65 have mild cognitive impairment (MCI), defined as experiencing more memory problems than normally expected with aging, but no other symptoms of dementia such as impaired judgment or reasoning. Persons with MCI (patients) are at great risk for developing dementia (10-33% per year). Memory problem (poor executive function) diminish the patient's confidence and ability to perform meaningful and/or important activities (e.g. socialization, medication management).

Deteriorating life satisfaction in patients and care partners (caregivers) is a prevalent problem due to diminished meaningful activity engagement which occurs as a result of patient frustration and embarrassment, lack of self-efficacy (confidence), and diminishing activity performance. As a result, patients experience additional negative health outcomes: 38% report depressive symptoms and anxiety. Caregivers often lack confidence to manage their own and the patient's daily challenges and meaningful activity engagement, leading to high caregiver burden, depressive symptoms, and anxiety. As a dyad, both patients and caregivers report diminished satisfaction within their communication and relationship due to disagreement about the patient's functional ability to effectively and safely perform meaningful activities.

Emerging evidence indicates regular engagement in social, physical or cognitive activities can improve life satisfaction, activity performance, depressive symptoms, anxiety, and dyad communication; health outcomes are even better when the activities are self-selected and meaningful. To promote patients' and caregivers' life satisfaction and health outcomes, interventions to maximize patients' capacity for full engagement in meaningful activities are essential; yet, there is a marked absence of such empirically validated interventions.

The investigators developed and tested the Daily Engagement in Meaningful Activities (DEMA) intervention to improve life satisfaction and health outcomes for patients and caregivers. DEMA is a positive health focused, theoretically grounded, tailored, family-centered, multi-faceted intervention. Over 7 session, dyads work with a nurse to 1) identify meaningful activities, assess capacity, problem-solve barriers, and establish routines for engagement and 2) learn more about MCI by working through six Self-Management Toolkit topics (e.g., benefits of meaningful activity; planning the future).

The investigators' purpose is to evaluate the efficacy of DEMA in a two-group randomized controlled trial with 200 patient/caregiver dyads (DEMA intervention vs. the information support (IS) attention control group).

Aim 1 (Primary Objective): Test DEMA's efficacy for improving life satisfaction in patients and their caregivers over time.

Aim 2 (Secondary Objective): Over time, evaluate DEMA's efficacy for patient and caregiver to:

1. increase patient activity performance and diminish depressive symptoms and anxiety.

   Hypothesis 2.1: Compared to the IS group, patients receiving DEMA will have improved activity performance and decreased depressive symptoms and anxiety.
2. decrease caregivers burden, depressive symptoms, and anxiety . Hypothesis 2.2: Compared to the IS group, caregivers receiving DEMA will have decreased burden, depressive symptoms, and anxiety.

Aim 3: Explore improvement in health outcomes over time in the sub-sample of patients with depressive symptoms using the (PHQ)-9 ≥ 5 at baseline) and explore the burden on caregivers when patients have PHQ-9 is >5. Compared to the non-depressed participants:

Hypothesis 3.1. Patients with depressive symptoms (scores > 5 on PHQ-9 measured at baseline) will have improved activity performance.

Hypothesis 3.2 Caregivers of patients with depressed symptoms (scores > 5 on PHQ-9 measured at baseline) will report reduced burden.

Hypotheses 3.3. Patients with depressive symptoms (scores > 5 on PHQ-9 measured at baseline) and their caregivers randomized to DEMA will report improved: confidence to manage daily challenges, communication satisfaction, life satisfaction, relationship satisfaction, decreased depressive symptoms and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Both the MCI patient and caregiver must consent to participate and have a phone at home or daily access to a telephone to be eligible for the study.

MCI patients will be eligible, if they:

* are aged > 59 years old;
* able to speak and read English;
* have both self or informant reported cognitive complaints,
* have MoCA score = 15 to 25
* are in the normal range in performance of daily living tasks based on functional impairment absent: a check box of Functional Activities Questionnaire (FAQ) has no score ≥2);

Family caregivers (spouse, other family members or friends) will be eligible, if they

* self-identify as care partner
* are aged ≥ 18 years old,
* have primary responsibility for providing unpaid care to an MCI patient, along with monitoring safety and providing social support;
* are able to speak and read English;
* are oriented to persons, places, and time (having a 6-item Screener score of 4 or above).

Exclusion Criteria:

* MCI patients and family caregivers will be excluded, if the MCI patient or family caregiver dyads participants are:

  * a diagnosed untreated severe major depression, or receiving advanced cancer treatment or hospice care,
  * receiving dialysis,
  * severe hearing loss and no hearing aids,
  * have no access to a telephone
  * the family caregiver has significant cognitive impairment that may hinder participation (6-item MMSE < 4).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Life satisfaction | Change from Baseline Life Satisfaction at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  The Life Satisfaction Index for the Third Age (LSITA) Scale-Short Form, is a 12-item with a 6-point response scale (ranging from "1" Strongly disagree to "6" strongly agree) (Barrett & Murk, 2006). It is a measure of the overall construct of Life Satisfaction. It has been commonly used in older populations. Possible range of total scores is 12-72 and higher scores indicate better functioning. The total score ranges from 12 to 72.The reliability of the LSITA-SF scale was .90 (Barrett & Murk, 2006). The scale takes about 3 minutes to complete it. The LSITA is completed by patient and caregiver separately.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 Items (PHQ-9) | Change from Baseline PHQ-9 at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  Patient Health Questionnaire-9 Items (PHQ-9) is used to measure emotional function (Kroenke, Spitzer, & Williams, 2001). The PHQ-9 contains nine questions about symptoms. It has been widely used in older populations. The depression severity levels are: The scores 0 -4 indicate none, the scores between 5 to 9 indicate mild depression; the score between 10-14 indicates moderate depression; the scores between 15 to 19 indicate moderately severe depression, the scores between 20 to 27 indicate severe depression. The internal reliability was 0.83 to 0.92 (Kroenke et al., 2001). The scale takes about 3 minutes to complete it. The PHQ-9 is completed by patient and caregiver separately.
The General Anxiety Disorder 7-item (GAD-7) | Change from Baseline GAD-7 at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  The General Anxiety Disorder 7-item (GAD-7), four-point Liker scale is used to measure emotional function and it contains 7 questions about anxiety (Spitzer, Kroenke, Williams, & Lowe, 2006). It has been widely used in older populations. The GAD-7 scale score ranges from 0 to 21 and high scores indicates perceiving high level of anxiety. The internal reliability was 0.92 and test-retest reliability was 0.83 (Spitzer et al., 2006). The scale takes about 3 minutes to complete it. The GAD-7is completed by patient and caregiver separately.
Alzheimer Disease Cooperative Study MCI-Activities of Daily Living Inventory [ADCS-MCI-ADL Scale] | Change from Baseline ADCS-MCI-ADL at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  The 23-item ADCS-MCI-ADL Scale has good test-retest reliability, will be utilized to assess performance functioning in MCI patients (Galasko et al., 1997; Douglas Galasko et al., 2006; Pedrosa et al., 2010). The ADCS-ADL includes 18 items from traditional basic ADL scales and 5 items from instrumental activities of daily living scales (IADL) The possible range of total scores for the ADL Scale is 0-53 and higher scores indicate better functioning. The internal reliability was .91( Galasko et al., 1997; Douglas Galasko et al., 2006; Pedrosa et al., 2010). The scale takes about 15 minutes to complete it.
Relationship Assessment Scale (RAS) | Change from Baseline RAS at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  The Relationship Assessment Scale is a 7-item, 5 points Likert scale designed to measure general relationship satisfaction (Graham, Kunik, Doody, & Snow, 2005). The RAS was produces more reliable scores when administered to older individuals, older relationship, and married couples but it was intended to be applicable to a wide range of relationship types (Graham et al., 2005). Respondents answer each item using a 5-point scale ranging from 1 (low satisfaction) to 5 (high satisfaction). The total score ranges from 7 to 35.The internal reliability was .86-.87. The scale takes about 3 minutes to complete it.
Caregiving Outcomes Scale (COS) | Change from Baseline COS at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  The Bakas Caregiving Outcomes Scale (COS), a 15-item with a 7-point scale, self-report inventory, will be utilized to assess family caregiver outcomes. The scale has been used in family caregivers of those with a variety of other chronic conditions (Bakas, Champion, Perkins, Farran, & Williams, 2006; Pressler, 2008). It is one of recommendation instruments that can be used to identify priority areas for nursing intervention designed to improve caregivers' outcomes (Bakas et al., 2006; Deeken, Taylor, Mangran, Yabroff, & Ingham, 2003). It includes caregiver's financial well-being, level of energy, role functioning, physical functioning, and general health. The internal consistency reliability was provided alpha = .90 (Bakas et al., 2006). The scale takes about 5 minutes to complete it.

OTHER OUTCOMES:
Confidence Scale | Change Baseline Confidence Scale at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  The Nowotny Confidence Subscale (NCS) of the Nowotny Hope Scale is a self-report of confidence in one's own ability, which uses a 4-point Likert response format of strongly agree to strongly disagree. Content validity was established by literature review and an expert panel (Nowotny, 1989). The total score ranges from 8 to 32 and a higher score indicates better sense of confidence. .Concurrent validity of the entire scale was established with the Beck Hopelessness Scale at r = -0.47. The internal reliability was 0.83 to 0.92 (Nowotny, 1989.) The scale takes about 3 minutes to complete it.
The subscale of Communication and Affective Responsiveness (CAR) | Change from Baseline subscale of CAR at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  The subscale of Communication and Affective Responsiveness of The Family Assessment Device (FAD) is a 12-item, self-report questionnaire with 4-point responses Likert Scale (from 1 = strongly disagree to 4 = strongly agree) (Miller, Epstein, Bishop, & Keitner, 1985). These scales will be used to measure the satisfaction with communication with family members. The total score ranges from 12 to 48.The internal reliability was .90 (Miller et al., 1985). The scale takes about 4 minutes to complete it.
Dementia Deficits Scale (DDS) (Patient vs. Caregiver Versions) | Change from Baseline DDS at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  The Dementia Deficits Scale (DDS), patient version is used to assess MCI patients' awareness of the performance capacity (Snow et al., 2004). This multidimensional scale measures memory, attention, orientation, language, executive functioning, emotional and behavioral symptoms, and functional abilities. The patient rates him or herself performance capacity. Items are coded "0" if the deficit or symptom is not present or "1" if the deficit/symptom is present. The total score ranges from 0 to 35. The internal reliability for DDS with patient version was 0.77 to 0.91(Snow et al., 2004). The scale takes about 12 minutes to complete it.
The Canadian Occupational Performance Measure (COPM) | Change from Baseline COPM at Session 1(at Week 1), Session 2(at Week 2), Session 3 (at Week 4), Session 4 (at Week 6), Session 5 (at Week 8), Session 6 (at Week 10); Session 7 (at Week 12), 10 days post-, 3 months post-, and 6 months-post intervention
  The Canadian Occupational Performance Measure (COPM)-Importance subscale will be used to assess MCI patient's meaningful daily activities (Law et al., 1994). It is a generic measure with a semi-structured interview in which the patient is encouraged to identify problems in self-care, productivity or leisure activities. It is a widely known and valuable tool to assist in client-centered physical activity intervention studies. It concerns those activities the patient wants, needs, or is expected to do, but cannot to do, or those in which the patient is not satisfied with current performance. Then the patients will rate importance of the problems on a 10-point scale from "Not important at all" to "extremely important" (score 10). The internal reliability was 0.86 to 0.95 (Law et al., 1994)
The modified Credibility/Expectancy Questionnaire (CEQ) | 10 days post-intervention evaluation
  The 6-item Credibility/Expectancy Questionnaire (CEQ) is used to assess participants (patient/caregivers) perception of intervention credibility/expectancy (Devilly & Borkovece, 2000). This multidimensional scale measures credibility and expectancy of intervention or program. The scale is from 1 to 9. The item coded 1 to 3 for "Not at all", 4 to 6 for Somewhat, or Very for 7 to 9. The items 1, 2, and 3 are loading on factor credibility; the items 4, 5, and 6 are loading on factor expectancy. The total score ranges from 1 to 42. The internal reliability of CEQ was 0.79 to 0.90 (Devilly & Borkovece, 2000). The scale takes about 3 minutes to complete it.
Six-item Screener [Completed by caregiver] | Pre-consent
  The six-item screener is a subset of the full MMSE, a brief cognitive screener with acceptable sensitivity (86%) and specificity (91%) for identifying subjects with cognitive impairment (Callahan, Unverzagt, Hui, Perkins, & Hendrie, 2002). It can be readily incorporated into an initial patient assessment of eligibility. The scale takes only 1 to 2 minutes to complete as compared with 7 to 15 minutes for longer scales. In addition, the six-item screener can be easily administered by telephone or in face-to-face interviews. The research can alter the cut-off score to match the goals of the study and the targeted population and diagnosing dementia using a cut-off score of 5 (range of possible scores 0-8 (Callahan et al., 2002). This measure has been used for identify family caregivers with cognitive impairment and it took only 2 minutes to complete it.
The Montreal Cognitive Assessment (MoCA) [Completed by Patient] | Pre-consent
  The Montreal Cognitive Assessment (MoCA) is a rapid screening instrument designed to help health professionals detect mild cognitive dysfunction (Nasreddine et al., 2003; Nasreddine et al., 2005). It assess numerous cognitive domains: attention and concentration, executive functions, memory, language, visuoconstrutional skills, conceptual thinking, calculation, and orientation. Time to administer is approximately 10 minutes. The total possible scores is 30 points; a score of 26 or above is considered normal. The test-reliability was .92 and the internal consistency was .83 ( Nasreddine et al., 2005). The high sensitivity of MoCA was found for identifying both AD and MCI patients (100% and 90%, respectively), specificity of the MoCA (defined as the ability to identify non-cognitively impaired subjects) was 87%. Positive and negative predictive values were also high for both AD patients (89% and 100%, respectively) and MCI patients (89% and 91%, respectively) (Nasreddine et al., 2005).
University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) [Completed by patients] | Pre-consent
  To further evaluate patient ability to provide informed consent, we will now use the 10-item (total score range 0-20) University of California, San Diego Brief Assessment of Capacity to Consent (UBACC):[23] internal consistency, Cronbach's ɑ = 0.77; interrater reliability, r = 0.44-0,73; concurrent validity acceptable, sensitivity (89%) and high specificity (100%);[23] and takes less 5 minutes to complete. Following a basic, verbal description of the study, potential patients will next complete the UBACC. The cut off point for patient self-consent is > to 14.
Demographic Profile and Comorbidity Condition | at Baseline, Pre-intervention Evaluation
  The demographic profile is completed by patient/caregiver and it has 32 items and includes MCI patient and caregiver demographic characteristics: recruitment setting, age, gender, education, relationship with patient, social economic status. Patient's MoCA scores and FAQ scores, and comorbidity condition (i.e. stroke, heart disease, or others). These are antecedent variables. Time to administer the Demographic Profile is Approximately.
Patient's Anti-depression medication and Anxiety Medication (Medication type, dosage, and using time frame) | Changes from Baseline patient's Anti-depression and Anxiety Medication at 10 days post-intervention evaluation, 3 months post-intervention, and 6 months post-intervention
  MCI patient/caregivers anti-depression medication and anti-anxiety medication information/using anti-depression/anti-anxiety medication or not (i.e., selective serotonin reuptake inhibitors [SSRIs]; Zoloft, Prozac, et al.)
Functional Activities Questionnaire (FAQ) [for MCI patient] | Pre-consent
  Functional Activities Questionnaire (FAQ) is, a 10-item, used to assess functional activities, which uses a 4-point Likert response format from "normal = 0" to "dependent = 3"(Mayo, 2016; Pfeffer, Kurosaki, Harrah, Chance, & Filos, 1982) The range of FAQ scores are from 0-30 and a cut-point of 9 (dependent in 3 or more activities) is recommended to indicate impaired function and possible cognitive impairment. The scale sensitivity is ranging from 85% to 98% and specificity ranging from 71% to 91% (Mayo, 2016; Pfeffer et al., 1982). Time to administer is approximately 5 minutes. FAQ is completed by patient or obtained from the medical record after receiving permission form the MCI patient. The FAQ has been used as part of the NIH Funded, Indiana Alzheimer Disease Center Uniform Data Set.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Y Lu, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Alzhemier Disease Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Roberts JL, Clare L. Meta-representational awareness in mild cognitive impairment: an interpretative phenomenological analysis. Aging Ment Health. 2013;17(3):300-9. doi: 10.1080/13607863.2012.732033. Epub 2012 Oct 16. PMID 23072638
- [Background] Plassman BL, Langa KM, McCammon RJ, Fisher GG, Potter GG, Burke JR, Steffens DC, Foster NL, Giordani B, Unverzagt FW, Welsh-Bohmer KA, Heeringa SG, Weir DR, Wallace RB. Incidence of dementia and cognitive impairment, not dementia in the United States. Ann Neurol. 2011 Sep;70(3):418-26. doi: 10.1002/ana.22362. Epub 2011 Mar 18. PMID 21425187
- [Background] Ward A, Tardiff S, Dye C, Arrighi HM. Rate of conversion from prodromal Alzheimer's disease to Alzheimer's dementia: a systematic review of the literature. Dement Geriatr Cogn Dis Extra. 2013 Sep 28;3(1):320-32. doi: 10.1159/000354370. eCollection 2013. PMID 24174927
- [Background] Apostolova LG, Cummings JL. Neuropsychiatric manifestations in mild cognitive impairment: a systematic review of the literature. Dement Geriatr Cogn Disord. 2008;25(2):115-26. doi: 10.1159/000112509. Epub 2007 Dec 14. PMID 18087152
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Pedrosa H, De Sa A, Guerreiro M, Maroco J, Simoes MR, Galasko D, de Mendonca A. Functional evaluation distinguishes MCI patients from healthy elderly people--the ADCS/MCI/ADL scale. J Nutr Health Aging. 2010 Oct;14(8):703-9. doi: 10.1007/s12603-010-0102-1. PMID 20922349
- [Background] Galasko D, Bennett D, Sano M, Ernesto C, Thomas R, Grundman M, Ferris S. An inventory to assess activities of daily living for clinical trials in Alzheimer's disease. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S33-9. PMID 9236950
- [Background] Galasko D, Bennett DA, Sano M, Marson D, Kaye J, Edland SD; Alzheimer's Disease Cooperative Study. ADCS Prevention Instrument Project: assessment of instrumental activities of daily living for community-dwelling elderly individuals in dementia prevention clinical trials. Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S152-69. doi: 10.1097/01.wad.0000213873.25053.2b. PMID 17135809
- [Background] Graham DP, Kunik ME, Doody R, Snow AL. Self-reported awareness of performance in dementia. Brain Res Cogn Brain Res. 2005 Sep;25(1):144-52. doi: 10.1016/j.cogbrainres.2005.05.001. PMID 15919186
- [Background] Bakas T, Champion V, Perkins SM, Farran CJ, Williams LS. Psychometric testing of the revised 15-item Bakas Caregiving Outcomes Scale. Nurs Res. 2006 Sep-Oct;55(5):346-55. doi: 10.1097/00006199-200609000-00007. PMID 16980835
- [Background] Pressler SJ. Cognitive functioning and chronic heart failure: a review of the literature (2002-July 2007). J Cardiovasc Nurs. 2008 May-Jun;23(3):239-49. doi: 10.1097/01.JCN.0000305096.09710.ec. PMID 18437066
- [Background] Deeken JF, Taylor KL, Mangan P, Yabroff KR, Ingham JM. Care for the caregivers: a review of self-report instruments developed to measure the burden, needs, and quality of life of informal caregivers. J Pain Symptom Manage. 2003 Oct;26(4):922-53. doi: 10.1016/s0885-3924(03)00327-0. PMID 14527761
- [Background] Nowotny ML. Assessment of hope in patients with cancer: development of an instrument. Oncol Nurs Forum. 1989 Jan-Feb;16(1):57-61. PMID 2911528
- [Background] Snow AL, Norris MP, Doody R, Molinari VA, Orengo CA, Kunik ME. Dementia Deficits Scale. Rating self-awareness of deficits. Alzheimer Dis Assoc Disord. 2004 Jan-Mar;18(1):22-31. doi: 10.1097/00002093-200401000-00005. PMID 15198084
- [Background] Law M, Polatajko H, Pollock N, McColl MA, Carswell A, Baptiste S. Pilot testing of the Canadian Occupational Performance Measure: clinical and measurement issues. Can J Occup Ther. 1994 Oct;61(4):191-7. doi: 10.1177/000841749406100403. PMID 10137673
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Callahan CM, Unverzagt FW, Hui SL, Perkins AJ, Hendrie HC. Six-item screener to identify cognitive impairment among potential subjects for clinical research. Med Care. 2002 Sep;40(9):771-81. doi: 10.1097/00005650-200209000-00007. PMID 12218768
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Jeste DV, Palmer BW, Appelbaum PS, Golshan S, Glorioso D, Dunn LB, Kim K, Meeks T, Kraemer HC. A new brief instrument for assessing decisional capacity for clinical research. Arch Gen Psychiatry. 2007 Aug;64(8):966-74. doi: 10.1001/archpsyc.64.8.966. PMID 17679641
- [Background] Pfeffer RI, Kurosaki TT, Harrah CH Jr, Chance JM, Filos S. Measurement of functional activities in older adults in the community. J Gerontol. 1982 May;37(3):323-9. doi: 10.1093/geronj/37.3.323. PMID 7069156

DOCUMENTS (1):
  • Informed Consent Form (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT04515875/ICF_000.pdf